CLINICAL TRIAL: NCT02448199
Title: Phase III Study Comparing Association of Anti-inflammatory and Anti-rheumatic
Brief Title: Study of Association of Anti-inflammatory and Anti-rheumatic
Acronym: ZDPC00213
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zodiac Produtos Farmaceuticos S.A. (Industry)
Collaborators: Eurotrials Brasil Consultores Cientificos Ltda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Zodiac Produtos Farmacêuticos
Record Dates: First submitted 2015-05-11; First posted 2015-05-19 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Osteoarthritis
Keywords: pain; Knee
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — Meloxicam; Glucosamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Kit 1 ( ML + CG ) + P (Experimental): One sachet meloxicam and glucosamine and 1 placebo tablet once a day for 12 weeks One sachet
  Interventions: Drug: Meloxicam and Glucosamine
- Kit 2 ( ML + P) (Active Comparator): One tablet of meloxicam and one sachet of placebo once per day for 12 weeks
  Interventions: Drug: Meloxicam
- Kit 3 ( P+ GC) (Active Comparator): One sachet of glucosamine and one tablet placebo once a day for 12 weeks
  Interventions: Drug: Glucosamine

INTERVENTIONS:
Drug: Meloxicam and Glucosamine — Experimental
  Other Names: Association Anti-inflamatory/Anti-rheumatic
  Arms: Kit 1 ( ML + CG ) + P
Drug: Meloxicam — Active Comparator
  Other Names: Anti-inflamatory/Placebo
  Arms: Kit 2 ( ML + P)
Drug: Glucosamine — Active Comparator
  Other Names: Anti-rheumatic/Placebo
  Arms: Kit 3 ( P+ GC)

SUMMARY:
Phase III Study, double-blind, comparing association of anti-inflammatory and anti-rheumatic in 375 subjects with knee osteoarthritis.

DETAILED DESCRIPTION:
Evaluation after 12 weeks of treatment, in 3 arms, the efficacy and safety of the association.

ELIGIBILITY:
Inclusion Criteria:

* Signs the Informed Consent Form
* Age between 40 and 85 years
* osteoarthritis of the knee according to clinical and radiological criteria of the American College of Rheumatology

Exclusion Criteria:

* Cardiovascular disease
* Serious chronic comorbidity
* Hypersensitivity to any component of the study drugs
* body mass index> 30 kg / m²

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy measured by decrease in score algofunctional Lequesne index after 12 weeks from the start of treatment | 12 weeks
  Decrease in score of algofunctional Lequesne index after 12 weeks from the start of treatment

SECONDARY OUTCOMES:
Safety measured by frequency of adverse event | 12 weeks
  Safety as measured by total frequency of adverse event during the 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Edio Costa, Doctor, Study Chair — CRM